CLINICAL TRIAL: NCT07254403
Title: Anabolic Response to Beef vs Plant Protein in (Pre)Frail Older Adults Using a Novel Stable Isotope Pulse Method
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Professor, Texas A&M University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 107-Beef
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Protein Metabolism
MeSH Terms: interventions — Red Meat; Soy Foods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Frail older adults (Experimental): based on the Fried index
  Interventions: Other: Beef; Other: Tofu; Other: Placebo
- Pre-Frail Older Adults (Experimental): based on the Fried index
  Interventions: Other: Beef; Other: Tofu; Other: Placebo
- Non-Frail Older Adults (Experimental): based on the Fried index
  Interventions: Other: Beef; Other: Tofu; Other: Placebo

INTERVENTIONS:
Other: Beef — Beef, ground, 93% lean meat / 7% fat, patty, cooked, broiled: 100g = 26.2 g protein
Other: Tofu — Fried tofu: 100g = 18.8 g protein
Other: Placebo — water (to correct the anabolic data obtained after intake of the proteins for baseline (postabsorptive) values

SUMMARY:
Frailty is a common clinical syndrome in older adults that increases the risk for poor health outcomes including falls, disability, hospitalization, and mortality. Previous research showed increased protein needs and reduced anabolic response to meals in older adults, indicating the need for proteins with a high anabolic capacity to prevent and attenuate physical and cognitive health decline throughout the frailty cycle. Recently, more people have chosen to eliminate animal (i.e., beef) products from their diets which is concerning because of beef's anabolic properties due to high essential amino acid (EAA) levels and many other positive health effects. The Researchers' recently developed stable isotope amino acid pulse method enables measurement of the true intracellular anabolic response to a meal and bioavailability of food-derived amino acids. The research objective is to examine differences in the anabolic response and bioavailability of individual EAA and non-essential amino acids (NEAA) in beef as compared to plant protein in older adults with and without (pre-)frailty.

DETAILED DESCRIPTION:
Beef protein is known for its anabolic properties due to its high EAA levels and digestibility (~ 94% compared to 78% in beans and 86% in whole wheat). However, whether beef has the most optimal composition of individual EAA and non-essential amino acids (NEAA) for older adults with (pre)frailty remains unclear as well as the role of the individual branched-chain amino acids (BCAA) leucine, isoleucine and valine. Research is of scientific and clinical importance to understand whether (pre)frail older adults respond better to certain protein sources (i.e., beef protein) due to a more optimal profile/pattern of individual EAA and NEAA amino acids.

The study will take place at the research facility of the Center for Translational Research on Aging and Longevity (CTRAL), Texas A&M University located in the Human Clinical Research Building ) affiliated with Texas A&M University. The study involves 1 screening visit of approx. 3 hours, and 4 study days. Some study procedures (e.g., body composition, skeletal muscle function, questionnaires) may be skipped if completed within the past 3 months at CTRAL. All data will be recorded in Case Report Form and stored in the Texas A&M REDCap System. Subjects will be asked to arrive in the fasted state on all study days. Fasting prior to screening is not required. On the screening day, body weight, height, and body composition by Dual-energy X-ray absorptiometry (DXA) will be measured. In addition, The Six-Minute Walk Test (6MWT) and skeletal muscle function tests will be assessed at the end of each screening visit. Each study visit will begin with vital signs. Before administration of the feeding or the tracer solution, baseline blood will be collected for measurement of the natural enrichment of metabolites. After the baseline sample is collected, feeding will begin and will be followed by tracers of several compounds that may be administered by IV pulse. Participants will receive bites and sips of nutrition every 20 minutes for 5 hours. Participants will consume, using a randomized cross-over design, using a bite feeding method of the following proteins: (1) beef, (2) tofu (soy as the most popular plant-based protein) or (3) water (placebo to correct the anabolic data obtained after intake of the proteins for baseline (postabsorptive) values).

ELIGIBILITY:
Inclusion criteria:

* Age 65-95 years old
* Ability to walk, sit down, and stand up (independently or with walking assistance device)
* No recent use (< 4 weeks prior to start of the study) of dietary supplements and medication influencing protein and amino acid metabolism (e.g., antibiotics, oral corticosteroids)
* Willingness to lay supine in bed for up to 6 hours
* Willingness and ability to comply with the protocol

Exclusion criteria

* Presence of malnutrition (BMI < 17 kg/m2), 2). BMI >35 kg/m2 to avoid weight-related metabolic disturbances,
* Established diagnosis and active treatment of chronic disease: Insulin-dependent diabetes mellitus, active malignancy, heart disease, kidney disease, liver disease, HIV/AIDS, Asthma (moderate to severe), Hep (A, B, or C)
* History of untreated metabolic disease including hepatic or renal disorder
* Presence of fever within the last 3 days
* Cirrhosis of liver
* Diagnosis of dementia, neurodegenerative disease (e.g., Alzheimer's disease, Parkinson's disease, Huntington's chorea, frontotemporal dementia).
* (Possible) pregnancy
* Presence of acute illness or metabolically unstable chronic illness
* Active dependence on alcohol or drugs
* Newly prescribed long-term oral corticosteroids
* Planned elective surgery requiring 2 or more days of hospitalization during the entire study
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject
* Already enrolled in another clinical trial
* Any condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient
* Known allergy to any of the components of the feeding (soy, beef)
* Established daily diet of vegetarian/vegan composition

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Protein and amino acid synthesis capacity of beef and soy protein in older adults measured by the use of stable isotope tracers | 6 weeks
  A novel stable isotope technique will be used to assess simultaneously the anabolic response and whole body production rates of a variety of amino acids to intake of both dietary proteins in sarcopenic older participants. The samples will be stored in laboratory freezers and the amino acid isotope enrichments and concentrations analyzed by Liquid Chromatography with tandem mass spectrometry (LC-MS/MS). The researchers will then conduct LC-MS/MS analysis, peak integration, calculation of amino acid concentrations and whole body productions from raw data.

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-06-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT07254403/ICF_000.pdf